CLINICAL TRIAL: NCT06108453
Title: A Drug-drug Interaction Study to Evaluate the Effect of Rifampicin on the Pharmacokinetics of Methotrexate in Elderly Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Chung, Jae Yong, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MRIE
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Drug Interactions
MeSH Terms: interventions — Methotrexate; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Experimental)
  Interventions: Drug: Methotrexate Sodium
- Methotrexate + Rifampicin (Experimental): Methotrexate + Rifampicin
  Interventions: Drug: Methotrexate Sodium; Drug: Rifampicin

INTERVENTIONS:
Drug: Methotrexate Sodium — Methotrexate oral administration alone
Drug: Rifampicin — Co-administration of methotrexate and rifampicin
  Arms: Methotrexate + Rifampicin

SUMMARY:
To investigate the effect of rifampicin on the pharmacokinetics of methotrexate.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy elderly volunteers aged 70 to 80 years at the time of screening visit
2. Those whose weight is between 50.0 kg and 90.0 kg and whose BMI (kg/m2) is between 18.0 and 30.0 at the time of screening visit

   ※ BMI(Body mass index) = Weight (kg) / {Height (m2)}
3. Those who are suitable as test subjects for this test as determined by the investigator through physical examination, clinical laboratory performance examination, and questionnaire, etc.
4. Those who voluntarily decided to participate and agreed in writing to follow the precautions after receiving a detailed explanation of this clinical trial and fully understanding it before the screening test

Exclusion Criteria:

1. Those with clinical evidence of significant respiratory, circulatory, kidney, gastrointestinal, liver, endocrine, blood, nerve (including ataxia), mental or other chronic diseases, alcohol or drug addiction within one year from the start date of the clinical trial (However, currently well-controlled hypertension, hyperlipidemia, arthritis, benign prostatic hyperplasia (mild), and cataracts (if surgery is performed) may be selected at the discretion of the investigator.)
2. Persons with a history of clinically significant hypersensitivity to clinical investigational drug ingredients or drugs containing ingredients of the same class, or other drugs (aspirin, antibiotics, etc.) or food
3. Those with a history of gastrointestinal disease (e.g. Crohn's disease, ulcer, etc.) or surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of the investigational drug
4. People with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
5. Those who showed the following results in the screening test:

   * Blood AST (SGOT), ALT (SGPT), total bilirubin: > 1.5 times the upper limit of normal range
   * WBC count < 3,500 /μL
   * eGFR (MDRD equation) < 60 mL/min/1.73 m2
6. Those who test positive for hepatitis B, hepatitis C, HIV, or syphilis in the screening test
7. Those with a history of drug abuse or who tested positive for drugs of abuse in a urine screening test
8. Those who drink alcohol continuously (exceeding 21 units/week, 1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking during the clinical trial period
9. Those who tested positive in the alcohol breath test at the time of the screening test
10. Those who are unable to stop smoking during the entire clinical trial period, starting from 3 months before the scheduled date of first administration of the investigational drug
11. Those who have taken drugs with known significant drug interactions or drugs that are deemed unsuitable by the investigator within 14 days of administering the investigational drug (however, those who can take a break from medication for 7 days before administration and during the hospitalization period are excluded)
12. Persons who cannot refrain from consuming foods containing St. John's Wort or grapefruit during the entire clinical trial period, starting 14 days before the scheduled date of first administration of the investigational drug.
13. Persons who have continuously consumed excessive caffeine (>5 units/day) or who cannot refrain from consuming caffeine/caffeine-containing foods (coffee, tea, nutrient tonic drink drinks, etc.) during the entire clinical trial period from 7 days prior to the scheduled date of first administration of the investigational drug
14. Those who have taken prescription drugs or herbal medicine within 2 weeks before the first administration date, or who have taken over-the-counter drugs (OTC) or health functional foods within 7 days (however, if other conditions are appropriate according to the judgment of the investigator, participation in the clinical trial can participate)
15. A person who has participated in a clinical trial targeting other healthy people within at least 6 months prior to conducting the relevant clinical trial
16. Those who have donated whole blood or component blood within 1 month within 2 months before the scheduled date of first administration of the investigational drug, or who have received a blood transfusion within 1 month
17. Persons judged by the investigator to be unsuitable for participation in this clinical trial due to clinical laboratory test results or other reasons

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-10-24 (Estimated); Study Completion 2024-11-24 (Estimated)

PRIMARY OUTCOMES:
Compare Cmax of methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2 Day 1)
  Compare the maximum concentration (Cmax) of methotrexate
Compare AUClast of methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2 Day 1)
  Compare the area under the plasma concentration-time curve to from 0 to last measurable time point (AUClast) of methotrexate
Compare AUCinf of methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2 Day 1)
  Compare area under the plasma concentration-time curve from 0 hours to infinite time (AUCinf) of methotrexate

SECONDARY OUTCOMES:
Compare Cmax of 7-hydroxy methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2 Day 1)
  Compare the maximum concentration (Cmax) of methotrexate
Compare AUClast of 7-hydroxy methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2 Day 1)
  Compare area under the plasma concentration-time curve to last measurable time point (AUClast) of 7-hydroxy methotrexate
Compare AUCinf of 7-hydroxy methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2 Day 1)
  Compare area under the plasma concentration-time curve from 0 hours to infinite time (AUCinf) of 7-hydroxy methotrexate

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea